CLINICAL TRIAL: NCT04681300
Title: Transcriptomic Landscape of T Lymphocytes of Atopic Dermatitis, Atopic Prurigo Nodularis (of Besnier) and Non-atopic Prurigo Nodularis (of Hyde) Using Single Cell RNA-sequencing
Acronym: PRURISEQ
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200325
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2020-12

CONDITIONS: Prurigo Nodularis; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with atopic Prurigo nodularis , non-atopic Prurigo nodularis or atopic dermatitis
  Interventions: Other: Skin biopsy
- Patients with plastic surgery interventions
  Interventions: Other: Plastic surgery remnants

INTERVENTIONS:
Other: Skin biopsy — a skin sample will be taken using a 4 mm punch biopsy in lesional skin
  Groups: Patients with atopic Prurigo nodularis , non-atopic Prurigo nodularis or atopic dermatitis
Other: Plastic surgery remnants — healthy skin from plastic surgery interventions
  Groups: Patients with plastic surgery interventions

SUMMARY:
Prurigo nodularis (PN) is a skin condition characterized by symmetrically distributed widespread, pruritic nodules that occurs in patients with chronic pruritus. There are 2 subtypes of PN depending on the association with an atopic dermatitis (AD) : atopic PN (Besnier) and non-atopic PN (Hyde). There are no approved therapies, and treatment options currently used have limited efficacy and their long-term use carries the risk of potential severe toxic effects.

The mechanisms triggering PN are still unknown. However, recent findings suggest a major role for the Th2 inflammatory pathway.

Beyond advancing the basic understanding of PN pathophysiology, our study might also pave the way for developing novel Th2-targeted therapeutic strategies for PN and AD. The primary objective of this study is to characterize the transcriptional profile of the T lymphocytes isolated from skin samples from patients with PN. This study will allow a gain a deeper understanding of the pathophysiologic mechanism of PN, a better classification of its subtypes, as well as their physiopathologic link with AD. Moreover, it will help shape new effective and safe therapeutic approaches in these diseases which are important for optimal therapeutic management.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years of age
* Signature of the written contentment
* Clinical diagnostic of PN defined by the following: a minimum of 20 PN lesions, in total on both legs, and/or both arms; an average worst itch score of ≥7. Atopic PN will be defined as PN associating clinical sings or history of AD according to Hanifin et Rajka criteria. Non-Atopic PN will be defined as PN non-associated with clinical sings or history of AD according to Hanifin et Rajka criteria.
* or confirmed diagnosis of AD according to Hanifin et Rajka criteria without associated PN.
* Washout period for topical treatments (> 1 week) ans systemic treatments (> 1 month).
* Indication and absence of contraindication to performing a skin biopsy as part of the treatment

Inclusion criteria for healthy controls:

* more than 18 years of age
* Signature of the written contentment
* Hospitalised in the plastic surgery department of Saint-Louis Hospital.
* No associated inflammatory or tumoral skin condition
* No contraindication for biopsy

Exclusion criteria :

* Presence of inflammatory or tumoral skin morbidities other than PN and atopic dermatitis
* Treatment induced pruritus
* Pruritus secondary to other medical conditions such as bullous dermatosis, renal insufficiency, infectious diseases, …)
* AD under biologic therapy
* Patient under guardianship or conservatorship
* No health insurance coverage
* Patient under State Medical Assistance (AME)
* Pregnancy or breastfeeding
* Persons deprived of their liberty by a judicial or administrative decision
* People undergoing psychiatric care making their consent impossible
* Adults who are the subject of a legal protection measure or unable to express their consent
* Patients unable to read and write

Exclusion criteria for healthy controls:

* Inflammatory or tumoral medical condition
* Biological therapy for any other medical condition
* Associated inflammatory or tumoral skin condition
* Pregnancy or breastfeeding
* Persons deprived of their liberty by a judicial or administrative decision
* People undergoing psychiatric care making their consent impossible
* Adults who are the subject of a legal protection measure or unable to express their consent
* Patients unable to read and write

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with confirmed diagnosis of atopic dermatitis (n=5), atopic prurigo nodularis (of Besnier) (n=5) and non-atopic prurigo nodularis (of Hyde) (n=5) or from surgical residues of normal skin (n=5).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
Transcriptional profile of the T lymphocytes | at inclusion

SECONDARY OUTCOMES:
Inflammatory pathways | at inclusion
Molecular differences | at inclusion

IPD SHARING:
Plan to Share IPD: Undecided